CLINICAL TRIAL: NCT05651815
Title: Graphene Photothermal Adjuvant Therapy for Mild Corona Virus Disease 2019: A Prospective Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Collaborators: Hohhot First Hospital (Unknown)
Responsible Party: Principal Investigator, Songqiao Liu, Zhongda Hospital, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2022075
Record Dates: First submitted 2022-11-28; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: Corona Virus Disease 2019; Randomized Control Trial; Adjuvant Therapy; Graphene Photothermal
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graphene adjuvant therapy combined with conventional therapy group (treatment group) (Experimental): Graphene adjuvant therapy combined with conventional therapy group (treatment group)：Contrasted to the control groups, the treatment groups will undergo 30-min of graphene adjuvant therapy every day for 7 d.
  Interventions: Device: Graphene spectrum light wave therapy room
- Conventional therapy group (control group) (No Intervention): Conventional therapy group (control group)：Patients will only receive the conventional treatment for COVID-19.

INTERVENTIONS:
Device: Graphene spectrum light wave therapy room — Undergo 30-min of graphene adjuvant therapy every day for 7 d.
  Arms: Graphene adjuvant therapy combined with conventional therapy group (treatment group)

SUMMARY:
This is a future-proof and randomized controlled clinical study on the clinical efficacy of graphene photothermal adjuvant therapy in Corona Virus Disease 2019(COVID-19) patients with mild symptoms. The objective is to examine the effect of graphene photothermal adjuvant therapy on the time line for such Corona Virus Disease 2019 patients to achieve a negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) nucleic acid test result, and their duration of disease. Patients who meet study criteria will be randomized into the Grapheme adjuvant therapy combined with conventional therapy group (treatment group) and the conventional therapy only group (control group). Contrasted to the control groups, the treatment groups will undergo 30-min of graphene adjuvant therapy every day for 7 d.

DETAILED DESCRIPTION:
Following enrollment, patients will be randomized into treatment or control groups. All groups will receive the same conventional therapy.

In addition, treatment groups will undergo Graphene adjuvant therapy 30 minutes per day for 7 d.

Upon completion of the treatment protocol, specific study endpoints will be compared between the treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for mild COVID-19.
* Patients aged 18-60 years (inclusive).
* No later than 48 h after testing positive and the onset of clinical symptoms
* Sign informed consent form.

Exclusion Criteria:

* Severe or critically patients with COVID-19.
* Resting heart rate over 120 beats per minute.
* Coronary heart disease patients with acute cardiac insufficiency.
* Acute exacerbation of chronic obstructive pulmonary disease（COPD）.
* Uncontrolled hypertension [resting systolic blood pressure(SBP) more than 180 mmHg and diastolic blood pressure(DBP) more than 90 mmHg]; uncontrolled diabetes(Random Plasma Glucose, RPG>16.7mmol/L, HbA1C>7.0%)
* Patients with severe cardiovascular, hepatic, renal and hematopoietic diseases.
* Pregnant or menstruating woman.
* Known or suspected history of active tuberculosis or extrapulmonary tuberculosis, patients with brucellosis, pneumonia-related illness from other causes
* COVID-19 patients for the second or more times
* Those who cannot cooperate due to various reasons
* Body temperature: more than 38℃.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The time from positive at baseline to negative SARS-CoV-2 nucleic acid test | through study completion, an average of 10 days
  The time for grouped patients to receive a negative SARS-CoV-2 nucleic acid test result, including both ORF gene Ct value≥35 and N gene Ct value≥35.

SECONDARY OUTCOMES:
Hospital stay | through study completion, an average of 15 days
  Time to hospitalization for COVID-19
Negative test rate within 7 days | 7 days
  the rate of negative test of patients
Mild to moderate rate within 14 days | 14 days
  Mild to moderate rate within 14 days

OTHER OUTCOMES:
Lymphocytes variation | through study completion, an average of 15 days
  Lymphocytes count

CONTACTS AND LOCATIONS:
Overall Officials: Songqiao Liu, PhD., Study Chair — Southeast University
Locations (1):
- Hohhot First Hospital, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No
We did not seek or receive approval for this data sharing from our Institutional Review Board .